CLINICAL TRIAL: NCT00567034
Title: Augmenting Zyprexa With Naltrexone: Normalization of the Weight Gain Side Effect and the CNS Reward and Sensory Function
Brief Title: Augmenting Zyprexa With Naltrexone to Ameliorate Metabolic Side-Effects
Acronym: Zyprexa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Igor Elman, MD, MD, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2006-P-0002381/3; F1D-US-X306
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Zyprexa; naltrexone; schizophrenia; Metabolic Syndrome; pain
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Metabolic Syndrome; Pain | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): taking naltrexone
  Interventions: Drug: naltrexone
- 2 (Placebo Comparator): taking placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: naltrexone — 50mg naltrexone, 1 tablet a day for 12 weeks.
  Arms: 1
Drug: placebo — lactose placebo, 1 capsule every day for 12 weeks
  Arms: 2

SUMMARY:
The main purpose of this study is to determine whether the opioid antagonist naltrexone is helpful in ameliorating the weight gain and other adverse metabolic side effects experienced by schizophrenic patients taking the second generation antipsychotic (SGA) Zyprexa. Schizophrenics may have an altered/enhanced endogenous opioidergic drive, and because of this, normally painful stimuli will be sensed as less painful in schizophrenics vs. healthy controls. A secondary hypothesis for this study is that naltrexone augmentation of Zyprexa will normalize subjective pain ratings. Our tertiary objective is to examine the safety and tolerability of naltrexone in Zyprexa-treated patients with schizophrenia.

DETAILED DESCRIPTION:
Zyprexa is one of the most commonly prescribed second generation antipsychotic drugs (SGAs), but its (and other SGA's) side effects contribute to the development of obesity and to the "Metabolic Syndrome." Both conditions, which are more prevalent even in unmedicated schizophrenic patients, are associated with increased cardiovascular morbidity and mortality. The mechanisms of these side effects are likely to be multifactorial and to involve peripheral and central factors alike. The present proposal asks a fundamental question: How the endogenous opioidergic systems are involved in Zyprexa-induced obesity and in related metabolic disturbances. We further hypothesize that if the excess of central opioid activity creates metabolic problems for patients, it is reasonable to expect amelioration of the symptoms through blockade of opioid receptors. The proposed project is designed to test this hypothesis by complimenting clinical psychopharmacology with pain medicine research and functional magnetic resonance imaging (fMRI) to empirically measure clinical outcomes of Zyprexa pharmacotherapy augmentation with the opioid receptor antagonist, naltrexone. Our objectives and hypotheses are as follows: to determine the effects of naltrexone on weight gain, metabolic (e.g., cholesterol, lipids, insulin, leptin and glucose levels), anthropometric and nutritional characteristics in Zyprexa treated schizophrenic patients, to examine the effects of naltrexone on subjective pain ratings, and to investigate the safety and tolerability of naltrexone in Zyprexa-treated schizophrenic patients.

ELIGIBILITY:
Inclusion Criteria:

* Meeting DSM-IV-TR criteria for schizophrenia/schizoaffective disorder, confirmed by clinical interview with PI and SCID-I.
* On a stable dose of Zyprexa (i.e., greater than or equal to 10mg/day and less than or equal to 30mg/day) for at least 2 months; patients on typical antipsychotics or in a medications-free state will be also included and used for baseline comparison.
* Sufficient clinical stability (i.e., BPRS psychotic symptoms score of less than 19; BPRS anxiety/depression symptoms score of less than 15).
* Participation approved by the treating psychiatrist.
* BMI greater than or equal to 30kg/m^2 or BMI greater than or equal to 27kg/m^2 plus one symptom of the "Metabolic Syndrome" (i.e., fasting blood sugar greater than 125mg/dL, hypertension or dyslipidemia).
* Sufficient social stability following study admission, such as having safe, reliable living quarters, telephone access and at least one living relative or significant other willing to assist the subject following discharge from the study and to assist the staff if necessary to locate the subject subsequently.
* English speaking and reading ability sufficient to comprehend consent without assistance.
* Good physical health, no history of significant medical, surgical, or neurological illness, including any history of head trauma.
* Right-handedness
* Able to cooperate and comply with study procedures.

Exclusion Criteria:

* DSM-IV-TR diagnosis of current drug/alcohol dependence.
* Any lifetime history of dementia, bipolar disorder, major depression, other psychotic disorder, past or current drug/alcohol dependence, past or current eating disorder.
* Potentially confounding neurological condition (e.g., seizure disorder, head trauma accompanied by loss of consciousness greater than ten minutes or amnesia, brain surgery, multiple sclerosis, Parkinson's disease), or potentially confounding medical condition (e.g., diabetes mellitus or other endocrinopathy, chronic obstructive pulmonary disease, congestive heart failure, hepatitis, hepatic failure or cirrhosis, AIDS, pacemaker, kidney problems, hypokalemia, edema, and allergy to glucose).
* Allergy or hypersensitivity to naltrexone
* Abnormal laboratory, ECG or EEG results, elevated serum aminotransferases.
* Use within the previous month of any potentially confounding medications such as opioid agonists (e.g., morphine or codeine) or drugs with prominent orexigenic/anorexigenic effects (e.g., anticholinergics), insulin, oral hypoglycemics, amphetamines, opioid analgesics, anti-depressants including tricyclics, MAO inhibitors or mirtazapine, as determined by history and/or urine toxicology screen.
* Patient is pregnant or planning on becoming pregnant.
* Any cognitive impairment that precludes informed consent.
* Any chronic pain condition and/or any condition that may require opioid treatment in the course of the study.
* Dangerousness: any suicidal, assaultive or homicidal risks

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-12; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Weight and Body Mass Index | 12 weeks

SECONDARY OUTCOMES:
Subjective pain ratings, fMRI activations in the a priori selected ROIs, waist, waist/hip ratio, fasting blood glucose, LDL cholesterol, HDL cholesterol, triglycerides, fat body mass, insulin, leptin, and food intake | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Igor Elman, M.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States